CLINICAL TRIAL: NCT00475696
Title: Long-Term Monitoring of Safety in Subjects Treated With Duloxetine for Bladder Overactivity
Brief Title: Urge Incontinence Bladder Overactivity Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6984; F1J-MC-SBBX
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2007-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine

SUMMARY:
Examine the efficacy and safety of duloxetine in subjects with symptoms of bladder overactivity due to pure detrusor instability or sensory urgency. Subjects in study will be permitted to escalate or de-escalate between 80 mg/day and 120 mg/day in consultation with the investigator and based on their adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Are female outpatients.
* Are at least 18 years of age.
* Are ambulatory and able to use a toilet independently and without difficulty.
* Have no language or cognitive barriers, agree to comply with the requirements of the protocol, and sign a written informed consent document prior to entry into the study.
* Are women of non-childbearing potential by reason of hysterectomy or natural menopause, or are women of childbearing potential agreeing to use a medically accepted means of contraception (for example, intrauterine device [IUD], oral or injectable contraceptives, implant, barrier device, sterilization, abstinence, or sex with a vasectomized male partner) for the duration of the study. Women using oral contraceptives or hormone replacement therapy must have a stable dose and regimen for 3 months prior to the study.
* Have post-void residual (PVR) volume 100 mL within 15 minutes of a spontaneous void.
* Patients must have predominant symptoms of bladder overactivity defined as meeting both of the following criteria:

  1. bothersome urinary urgency (the sensation of the urgent need to void for fear of leakage) for a minimum of 3 consecutive months prior to study entry, or urge urinary incontinence (UUI; the involuntary loss of urine preceded by urgency) for a minimum of 3 consecutive months prior to study entry
  2. abnormal frequency of micturition (an average voiding interval of 2 hours or less [2] during waking hours) as confirmed by at least two days of recording on the screening dairy collected at Visit 1.
* Have UDS established DI or sensory urgency (determined at Visit 2).
* Have responded appropriately to all screening questions prior to Visit 1.

Exclusion Criteria:

* Use any medication other than duloxetine for urinary incontinence within 1 day prior to starting study medication or at any time during the study.
* Use monoamine oxidase inhibitors (MAOIs) or other excluded medications within 14 days prior to starting study medication or at any time during the study.
* Have any of the following:

  * A significant arrhythmia despite antiarrhythmic medication, uncontrolled angina, or a significant abnormality on ECG within 6 months prior to study entry that, in the opinion of the investigator, requires investigation or intervention.
  * Any active cardiac ischemic condition, including myocardial infarction within 6 months prior to study entry
  * Uncontrolled or poorly controlled hypertension
  * Active seizure disorder
  * Unstable diabetes mellitus
  * Spinal cord lesions, multiple sclerosis, or other neurological abnormalities that affect the lower urinary tract
  * History of severe allergies requiring emergency medical treatment or multiple adverse drug reactions
  * History of chronic lung disease associated with four (4) or more acute exacerbations per year resulting in severe coughing
  * Active or chronic hepatitis A, B, or C.
* Are pregnant, have been pregnant in the previous 6 months, or have not resumed normal menstruation for 3 months prior to study entry due to breastfeeding.
* Are breastfeeding.
* Have received treatment within the last 30 days with a drug other than duloxetine that has not received regulatory approval in any country for any indication at the time of study entry.
* Have any condition, limitation, disease, or abnormal laboratory value that could, in the judgment of the investigator, preclude evaluation of response to duloxetine.
* Are directly affiliated with the conduct of this study, or are immediate family of someone directly affiliated with the conduct of this study (that is, Lilly employees, investigators, site personnel, or their immediate families). Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-11; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
To monitor the safety of duloxetine 80 mg/day-120 mg/day in women with bladder overactivity due to pure detrusor instability or sensory urgency.

SECONDARY OUTCOMES:
To assess the subject's self-perceived improvement since starting study medication as measured by change from baseline on the following validated 7-point scale, Patient's Global Impressions of Improvement scale (PGI-I).

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana, United States
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Townsville, Queensland, Australia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North York, Ontario, Canada

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com